CLINICAL TRIAL: NCT01649921
Title: The Effects of Interferon-gamma on Sepsis-induced Immunoparalysis, a Randomised Double-blind Placebo-controlled Pilot (Phase IIIb) Study
Brief Title: The Effects of Interferon-gamma on Sepsis-induced Immunoparalysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFN_sepsis
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2014-04

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; SIRS; Septic shock; Immunoparalysis; Interferon-gamma
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Interferon-gamma; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interferon-gamma (Active Comparator)
  Interventions: Drug: Interferon-gamma, Recombinant
- Saline 0.9% (Placebo Comparator)
  Interventions: Other: Saline 0.9%

INTERVENTIONS:
Drug: Interferon-gamma, Recombinant — Interferon-gamma (Immukine, Boehringer-Ingelheim, Alkmaar, the Netherlands), 100mcg subcutaneously, on days 0-2-4-7-9-11. Interferon-gamma treatment will be initiated when the noradrenalin dose is reduced to 50% of maximum dose, ensuring that the sepsis-induced pro-inflammatory phase has passed
  Arms: Interferon-gamma
Other: Saline 0.9% — subcutaneous administration on days 0, 2, 4, 7, 9, and 11.
  Arms: Saline 0.9%

SUMMARY:
The primary aim of this study is to assess the effects of adjunctive therapy with Interferon (IFN)-gamma on immune function in patients with septic shock in a placebo-controlled manner. Moreover, the investigators want to evaluate new markers that could be used to identify patients with immunoparalysis, and to monitor the patient's immunological response to IFN-γ. In addition, mechanistic studies will be performed to further elucidate mechanisms (such as epigenetic modifications) behind immunoparalysis and the effects of IFN-γ on these mechanisms. With use of the results the investigators will obtain in this pilot study, the investigators will conduct a large multicentre clinical trial with IFN-γ.

DETAILED DESCRIPTION:
Sepsis is the leading cause of death in the ICU with an estimated 6 million victims per year worldwide. Although septic shock is traditionally viewed as an excessive systemic inflammatory reaction to invasive microbial pathogens, pharmacological suppression of the innate immune response in sepsis has proved to be unsuccessful. An important reason for this might be that the vast majority of septic patients survive the initial pro-inflammatory hit, but die in the subsequent immunosuppressed state due to secondary/opportunistic infections. This so-called 'immunoparalysis' is increasingly recognized as the overriding immune dysfunction in septic patients. Reversal of sepsis-induced immunoparalysis is therefore a promising adjunctive treatment for patients presenting with septic shock.

It was demonstrated that interferon-gamma (IFN)-gamma can reverse immunoparalysis in vitro and in vivo in animals and in healthy volunteers. Moreover, in a case-series of septic patients interferon-gamma treatment leaded to reversal of immunoparalysis, reduction in mechanical ventilation time and length of stay with no relevant side-effects.

The primary aim of this study is to assess the effects of adjunctive therapy with IFN-gamma on immune function in patients with septic shock in a placebo-controlled manner. Moreover, the investigators want to evaluate new markers that could be used to identify patients with immunoparalysis, and to monitor the patient's immunological response to IFN-γ. In addition, mechanistic studies will be performed to further elucidate mechanisms (such as epigenetic modifications) behind immunoparalysis and the effects of IFN-γ on these mechanisms.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent from patient of legal representative
* Age >18 years
* Presence of septic shock of bacterial origin with evidence of bacterial infection (last 96 hours, with at least one pathogenic microorganism in blood, sputum, urine, normally sterile body fluid, or on central venous catheter; Focus of infection identified (e.g. ruptured bowel, purulent drainage/sputum); or leukocytes in normally sterile body fluid), Two SIRS criteria (last 24 hours, fever (>38.3 ˚C), hypothermia (<35.6 ˚C), tachycardia (>90bpm), tachypnea (>20/min), or partial pressure of arterial carbon dioxide (PaCO2) <32 mmHg, or mechanical ventilation, leukocytosis (>12,000/μl), leucopenia (<4,0000/μl), or >10% immature forms), and presence of shock with need for vasopressor therapy to maintain systolic blood pressure (SBP) ≥ 90 mmHg.

Exclusion Criteria:

* Pregnancy or lactating
* Subjects with a history of allergy or intolerance to IFN-gamma
* Systemic autoimmune disease, hematologic disease (neoplasma, acute leukemia), transplant patients, or patients on steroid medication receiving a prednisolone equivalent of > 5 mg per day
* Human immunodeficiency virus positivity
* Presence of an advanced directive to withhold or to withdraw life sustaining treatment
* Underlying disease with a prognosis for survival < 3 months, or moribund patient highly likely to die within 24 hours.
* Cardiopulmonary resuscitation (<72 hours) before enrollment
* Acute myocardial infarction or pulmonary embolization (<72 hours)
* Participation in a clinical trial until 30 days prior to inclusion
* Subjects with a history of documented epileptic seizures
* Subjects with severe renal impairment (creatinine clearance less than 30 mL/min)
* Subjects with severe liver failure (impaired synthesis of proteins such as coagulation factors manifested by increased prothrombin time)
* Subjects with an absolute neutrophil count of less than 500/mm3 at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the tumor necrosis factor (TNF)-α secretion by ex vivo lipopolysaccharide (LPS)-stimulated leukocytes as a marker of immunosufficiency/antimicrobial response. | at admission and at days 0, 2, 7, 14 and 28

SECONDARY OUTCOMES:
Outcome of bacterial infection (occurrence of secondary and/or opportunistic infections, duration of antibacterial treatment, microbiological evaluation) | At days 0, 2, 7, 14 and 28
Hemodynamic stability (noradrenalin infusion rate, amount of infused fluids per day, amount of urine produced per day, daily fluid balance) | At days 0, 2, 7, 14 and 28
Mortality (including time to death) at week 2 and week 6 after end of treatment (all causes) | At days 14 and 28
Length of stay at ICU and duration of hospitalization | At days 28 and 56
Organ function | at days 0, 14, and 28
  * Cardiovascular function: lactate level, vasopressor usage, and cardiovascular Sequential Organ Failure Assessment (SOFA) score
  * Respiratory function: oxygenation index, Pulmonary Arterial Oxygen Tension (PaO2) / fraction of inspired oxygen (FiO2) (P/F) ratio, and respiratory SOFA score
  * Renal function: creatinine level, urine output, renal replacement therapy usage, and renal SOFA score
  * Hematologic function: hematologic SOFA score
  * Hepatic function: Hepatic SOFA score
Production of other cytokines by leukocytes ex vivo stimulated with various stimuli (including LPS, peptidoglycan, candida) | At admission, at days 0, 2, 7, 14, and 28
Markers of "immune status" (including human leukocyte antigen expression on monocytes (mHLA)-DR and programmed death (PD)-1 expression, interleukin (IL)-6 plasma concentration) | At admission and at days 0, 2, 7, 14, and 28
the correlation between the level of immunoparalysis (indicated by the commonly used marker mHLA-DR and new markers of "immune status" found), and effectiveness of IFN-γ (indicated by TNF-α secretion by ex vivo LPS-stimulated PBMC's). | At days 0, 14, and 28
Transcriptional activity of leukocytes, including microarrays with a focus on inflammatory pathways | At admission and at days 0, 2, 7, 14, and 28
Changes in phenotype or gene expression caused by mechanisms other than changes in the underlying DNA sequence (epigenetic modifications) | At admission and at days 0, 7, and 28
reversibility of monocytes tolerance | Day 0
  the reversibility of monocytes tolerance by the mean of innate immune training (cytokines production such as TNF and Interleukin (IL)-6 will be assessed).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands